CLINICAL TRIAL: NCT05677230
Title: To Compare the Safety and Efficacy of Balloon Occluded/Plug Assisted Retrograde Transvenous Obliteration With Endoscopic Variceal Obturation for Primary Prophylaxis of Gastric Varices With Large Spontaneous Shunt: A Randomized Controlled Trial
Brief Title: To Compare the Safety and Efficacy of Balloon Occluded/Plug Assisted Retrograde Transvenous Obliteration With Endoscopic Variceal Obturation for Primary Prophylaxis of Gastric Varices With Large Spontaneous Shunt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-52
Record Dates: First submitted 2023-01-03; First posted 2023-01-10 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-08

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balloon Occluded/plug assisted Retrograde Transvenous Obliteration. (Experimental): Balloon occluded/plug assisted retrograde transvenous obliteration will be done one time only.
  Interventions: Procedure: Balloon occluded/plug assisted retrograde transvenous obliteration.
- Endoscopic Variceal Obturation (Active Comparator): endoscopic variceal glue therapy will be done till obturation every 3 weekly.
  Interventions: Procedure: Endoscopic Variceal Obturation

INTERVENTIONS:
Procedure: Balloon occluded/plug assisted retrograde transvenous obliteration. — Balloon occluded/plug assisted retrograde transvenous obliteration will be done one time only.
  Arms: Balloon Occluded/plug assisted Retrograde Transvenous Obliteration.
Procedure: Endoscopic Variceal Obturation — Endoscopic Variceal Glue Therapy will be done till obturation every 3 weekly.
  Arms: Endoscopic Variceal Obturation

SUMMARY:
Study population: All the consecutive patients of cirrhosis who are diagnosed to have large gastric varices without prior history of bleeding from GV, who came to OPD or endoscopy in Hepatology department of ILBS will be evaluated for inclusion.

Study design: Prospective interventional study. The study will be conducted in the Department of Hepatology ILBS.

Study period: 1.0 years

Sample size: 42

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Cirrhotic patients, with GV (GOV2 or IGV1) with eradicated or small low risk esophageal varices with gastrorenal shunt of >10 mm size amenable for BRTO/PARTO.

Exclusion Criteria:

1. Non-cirrhotic portal hypertension,
2. History of bleeding from GV
3. Hepatic encephalopathy grade III/IV,
4. Acute kidney injury
5. Patients on beta blocker therapy for > 6 months prior to enrollment in study
6. Hepatocellular carcinoma
7. Portal venous thrombosis
8. Presence of jaundice (bilirubin >3 mg/dl), ascites, Child C, MELD > 18
9. Advanced cardiac or pulmonary diseases
10. Pregnancy
11. Patients not giving informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patient having bleeding from GV at 12 months | 6 months

SECONDARY OUTCOMES:
Proportion of patients achieving complete or partial obturation of GV | 6 months
Proportion of patients having change in grade of EV and bleeding from EV | 6 months
Proportion of patients having appearance or worsening of PHG | 6 months
Change in HVPG in those patients who bleed after BRTO/PRTO | 6 months
Change in HVPG in those patients who bleed after EVO | 6 months
Change in liver (in KPa) and splenic stiffness (in KPa) after BRTO/PRTO using transient elastography | 6 months
Change in liver (in KPa) and splenic stiffness (in KPa) after using transient elastography | 6 months
Proportion of patients having new onset decompensation with ascites, jaundice or hepatic encephalopathy | 6 months
Proportion of patient developing post procedure liver failure | 6 months
Proportion of patient developing post acute kidney injury or sepsis | 6 months
Duration of hospital stay poof procedure | 12 months
Evaluation of expertise of endoscopists | 12 months
Any variceal bleed | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided